CLINICAL TRIAL: NCT02602041
Title: Knowledge and Attitudes Regarding Healthy Lifestyle and Health Behavior Change in Cancer Patients and Their Partners
Brief Title: Knowledge and Attitudes Regarding Healthy Lifestyle and Health Behavior Change in Cancer Patients and Their Partners; A Pilot Study
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 201501074
Record Dates: First submitted 2015-11-03; First posted 2015-11-11 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Testicular Cancer
MeSH Terms: conditions — Breast Neoplasms; Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with breast cancer and partners: We will invite 10 women with early stage breast cancer (BC) and their partners for a semi-structured interview.
  Interventions: Other: Literature search and semi-structured interview
- Patients with testicular cancer and partners: We will invite 10 men with disseminated testicular cancer (TC) and their partners for a semi-structured interview.
  Interventions: Other: Literature search and semi-structured interview

INTERVENTIONS:
Other: Literature search and semi-structured interview — We will do a literature search and perform semi-structured interviews with cancer patients and their partners in order to explore knowledge, attitudes, barriers and facilitators regarding health behavior change following cancer treatment.

SUMMARY:
The investigators will perform a pilot study to gain insight into attitudes, barriers and facilitators for health behavior change in cancer patients and their partners. Results of this pilot will be used to design suitable questionnaires to investigate health behavior change in a larger cohort of patients and their partners. It will also direct future interventions to adequately target patients and, potentially, their partners to improve their lifestyle following a cancer diagnosis.

DETAILED DESCRIPTION:
The investigators will perform semi-structured interviews with cancer patients and their partners in order to explore knowledge, attitudes, barriers and facilitators regarding health behavior change following cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 65 years of age
* have completed adjuvant or curative chemotherapy (in BC and TC patients, respectively) or started adjuvant hormonal therapy alone (in BC patients) between 6 and 24 months previously
* have no signs or symptoms of recurrent disease
* be in follow-up at the Department of Medical Oncology of the UMCG.

Exclusion Criteria:

* signs or symptoms of recurrent disease
* mental disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will invite 10 women with early stage breast cancer (BC) and 10 men with disseminated testicular cancer (TC) and their partners (20 couples in total).
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Gain insight into barriers and facilitators for health behavior change | 12 months
  Qualitative description of barriers and facilitators for health behavior change

CONTACTS AND LOCATIONS:
Overall Officials: J. Nuver, MD, PHD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands